CLINICAL TRIAL: NCT06584084
Title: Technical and Clinical Validation Study of a New Wireless Portable and Multi-Channel Surface EMG Device to Analyse Motor Unit Action Potentials
Brief Title: Technical and Clinical Validation of the WPM-SEMG Prototype
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alain Kaelin (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Alain Kaelin, Prof., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SUPSI-2017-006
Record Dates: First submitted 2018-01-23; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neuron Disease, Motor
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Each participant will undergo to the study intervention and the control intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle electrophysiological signals recording (Experimental): Recording of electrophysiological signals of muscles with a WPM-SEMG prototype
  Interventions: Device: WPM-SEMG prototype

INTERVENTIONS:
Device: WPM-SEMG prototype — Measurements will be done with the rigid matrix. The flexible electrode matrix will be used only on a lower percentage of volunteers depending on the results obtained with the rigid matrix

SUMMARY:
Validation study designed to demonstrate the technical and clinical performance, and the safety of a new medical device in healthy volunteers and patients with myopathy or neuropathy. The medical device is the WPM-SEMG prototype designed for recording electrophysiological signals of muscles.

DETAILED DESCRIPTION:
The study consists of two parts:

* the first part concerns the technical validation of the prototype. It will enrol 10 healthy volunteers (Technical Validation Group).
* the second part concerns the clinical validation of the prototype in comparison with the gold standard, that is the needle-EMG. It will enrol 50 healthy volunteers (Clinical Validation Group), including also the 10 subjects of the Technical Validation Group, and 20 patients

Measurements will be done on 4 muscles with the WPM-SEMG device prototype using a rigid electrode matrix. For each muscle, the participant will execute some spontaneous motor activities and measurements will be taken on the muscle under tension (low, medium, and high) for a total of 12 measurements. Measurements will be repeated two times after a pause for a total of 24 acquisitions. For the group with myopathies an additional fifth muscle, not foreseen by the protocol, can be done if considered the clinical most affected muscle followingthe neurological examination.

A control intervention is done on the same subjects and consists in a needle-EMG which will be applied as for routine clinical practice on the same muscles used for the WPM-SEMG device prototype. Measurements will be taken for each muscles as for the rigid matrix.

ELIGIBILITY:
Eligibility criteria for healthy volunteers

* Inclusion Criteria

  * Healthy volunteers
  * Female or male
  * 18 years or older
  * Preserved cognitive capacity
  * Ability to understand the study
  * Willingness to complete all the study assessments
  * No chronic or concomitant use of medications or treatment
  * Written informed consent
* Exclusion Criteria

  * Skin lesions in the area below the electrode
  * Allergy to metal alloys
  * History of skin disease
  * Pregnancy
  * Lactation
  * Known causes of neuromuscular disease
  * Inability to follow the procedures of the study

Eligibility criteria for patients

* Inclusion Criteria

  * Patients of the Neurocentro della Svizzera Italiana with diagnosis of myopathy or neuropathy that requires a needle-EMG electrophysiological testing as standard clinical management of the disease
  * Female or male
  * 18 years or older
  * Preserved cognitive capacity
  * Ability to understand the study
  * Willingness to complete all the study assessments
  * No chronic or concomitant use of medications or treatment that may influence the measure in the opinion of the investigator (muscle relaxant such as baclofen, statin, benzodiazepine).
  * Written informed consent
* Exclusion Criteria

  * Skin lesions in the area below the electrode
  * Allergy to metal alloys
  * History of skin disease
  * Cognitive and/or psychiatric disorders
  * Pregnancy
  * Lactation
  * Neuromuscular disease other than myopathy and neuropathy
  * Inability to follow the procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Technical and clinical assessment | Intervention (day0)
  Correlation between the properties of the final electrophysiological output identified from sEMG signals acquired with the WPM-SEMG device prototype and the properties of the final electrophysiological output identified from EMG signals acquired using needle EMG. [Time Frame: Intervention (day0)]
  The following properties will be extracted: Amplitude (microVolts), phases/turns (ratio), signal frequency (Hz) and duration (seconds).

SECONDARY OUTCOMES:
Pain assessment | Intervention (day0)
  Pain assessment during the measurements using the Visual Analog Scale (VAS). The VAS consists on a 0-10 scale, with two end points representing 0 ('no pain') and 10 ('worst possible pain').

CONTACTS AND LOCATIONS:
Locations (1):
- Neurocentro della Svizzera Italiana, Lugano, Switzerland